CLINICAL TRIAL: NCT04354220
Title: Accuracy of Capnography Monitoring in Invasively and Non-invasively Ventilated Children
Brief Title: Capnography Monitoring in Ventilated Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vincenzo Cannizzaro (Other)
Responsible Party: Sponsor-Investigator, Vincenzo Cannizzaro, Senior consultant and head of research, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: KISPI-CAPNO
Record Dates: First submitted 2019-04-16; First posted 2020-04-21 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Child, Only; Infant, Newborn, Diseases; Critical Illness; ARDS, Human; Heart Defects, Congenital; Lung Diseases, Obstructive; Lung Diseases, Interstitial
Keywords: capnography; end-tidal CO2; critically ill children; ventilated; accuracy
MeSH Terms: conditions — Infant, Newborn, Diseases; Critical Illness; Respiratory Distress Syndrome; Heart Defects, Congenital; Lung Diseases, Obstructive; Lung Diseases, Interstitial | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- no shunt, no lung injury: ventilated newborns / infants / children with healthy lungs and without or corrected congenital heart disease and no intra-/extra-cardiac shunt
  Interventions: Diagnostic Test: capnography monitoring; Diagnostic Test: arterial blood gas
- mild lung injury: ventilated newborns / infants / children with mild lung injury (OI between 4 and 8)
  Interventions: Diagnostic Test: capnography monitoring; Diagnostic Test: arterial blood gas
- moderate-severe lung injury: ventilated newborns / infants / children with moderate or severe lung injury (OI above 8)
  Interventions: Diagnostic Test: capnography monitoring; Diagnostic Test: arterial blood gas
- shunt lesion: ventilated newborns / infants / children with cyanotic heart diseases and therefore existing intra-cardiac or extra- cardiac right-left shunt lesions
  Interventions: Diagnostic Test: capnography monitoring; Diagnostic Test: arterial blood gas

INTERVENTIONS:
Diagnostic Test: capnography monitoring — routinely used capnography monitoring
Diagnostic Test: arterial blood gas — Routinely taken arterial blood gas values

SUMMARY:
End-tidal CO2 measurements in children will be assessed for their accuracy with arterial CO2 measurements.

DETAILED DESCRIPTION:
End-tidal and arterial CO2 measurements will be performed in invasively and non-invasively ventilated critically ill children. The endtidal CO2 values will assessed for their accuracy with respect to different underlying diseases and conditions of the children.

ELIGIBILITY:
Inclusion Criteria:

* Children on pressure controlled mechanical invasive or non-invasive ventilation on the Paediatric Intensive Care Unit of the University Children's Hospital Zurich
* Newborns with a birthweight of at least 2.0 kg
* Newborns with an age of at least 1 hour (age > 60 minutes)
* Children up to the last day of the 13th year of living
* Ability of care taker or patient to understand verbal and written instructions and the general consent or informed consent in German or English
* Obtained written general or informed consent as documented by signature
* Available arterial line, i.e. a specific catheter inserted in an artery

Exclusion Criteria:

* Care taker or participant unable for linguistic, mental or other reasons or unwilling to understand verbal or written information and to give written informed consent in German or English
* Care taker not available
* Newborns with a birthweight below 2.0 kg
* Newborns younger than 1 hour (age <60 minutes)
* Children with an age of 14 years onwards
* Missing arterial line
* Patients dependent on any other kind of respiratory support that is not compatible with the PcCO2-sensor or where a high leakage in the respiratory circuit makes PcCO2 measurements impossible (nasal mask ventilation, low-flow-/high-flow-ventilation, rebreathing mask, high- frequency-oscillation)
* Patients where the investigators act on the assumption that mechanical ventilation will be discontinued and/or the arterial line will be removed within 6 hours or where only one pair of values (arterial and endtidal CO2) can be compared
* Patients with a cyanotic shunt lesion with a weight of 15 kg or above

Ages: 1 Hour to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Critically ill infants and children under invasive and non-invasive mechanical ventilation, regardless of their underlying acute or chronic diseases, as long as an arterial line for blood gas analyses is in situ.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of end-tidal Carbon Dioxide (PetCO2) values in comparison to arterial Carbon Dioxide (PaCO2) values in invasively and non-invasively ventilated critically ill children without lung or heart disease | On average every participant will be assessed for 5 days
  Mean absolute measurement difference between simultaneously obtained PaCO2 and PetCO2 values (bias) and their 95% limits of agreement (precision) in children and newborns without cardiopulmonary dysfunction. Units of measure will be in kilopascal (kPa) for PetCO2 and PaCO2, respectively.

SECONDARY OUTCOMES:
Accuracy of end-tidal Carbon Dioxide (PetCO2) values in comparison to arterial Carbon Dioxide (PaCO2) values in invasively and non-invasively ventilated critically ill children with lung and or heart disease | On average every participant will be assessed for 5 days
  Cardiopulmonary function-dependent mean absolute measurement difference between simultaneously obtained PaCO2 and PetCO2 values (bias) and their 95% limits of agreement (precision) in children and newborns with cardiopulmonary dysfunction. Units of measure will be in kilopascal (kPa) for PetCO2 and PaCO2, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No